CLINICAL TRIAL: NCT02676193
Title: Effect of Packaging on Smoking Perceptions and Behavior: A Randomized Trial
Brief Title: Effect of Packaging on Smoking Perceptions and Behavior
Acronym: CASA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, David Strong, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R01CA190347 (NIH)
Record Dates: First submitted 2016-01-28; First posted 2016-02-08 (Estimated); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Smoking; Tobacco Smoking
Keywords: Tobacco Smoking; Cigarettes; Packaging; Text messaging; Graphic Images; Sensor-Based Assessments
MeSH Terms: conditions — Smoking; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Australian Packs (Experimental): The intervention to be administered to participants randomized to this group is the purchase of their US brand of cigarettes packaged using standard Australian marketing for three months.
  Interventions: Behavioral: Effect of Packaging on Smoking Perceptions and Behavior
- Blank Packs (Experimental): The intervention to be administered to participants randomized to this group is the purchase of their US brand of cigarettes packaged using blank packaging for three months. Blank packaging will indicate participants brand and will not have any brand-related images or labels.
  Interventions: Behavioral: Effect of Packaging on Smoking Perceptions and Behavior
- American Packs (No Intervention): Participants assigned the nonintervention group will purchase their US brand of cigarettes in the standard American packaging for three months.

INTERVENTIONS:
Behavioral: Effect of Packaging on Smoking Perceptions and Behavior — The intervention is the use of the assigned pack design.
  Arms: Australian Packs; Blank Packs

SUMMARY:
The investigators are addressing two critical areas identified by the FDA: the impact of cigarette packaging and labeling on consumer perceptions and on smoking behavior; and the effectiveness of graphic warning labels on communicating risk of tobacco products. In a randomized controlled trial (RCT), investigators will enroll committed smokers who have no intention of quitting in the next 6-months. The three study arms will be: a) a blank pack with all marketing materials removed (PP); b) The Australian graphic warning images (Australian model-AM); or c) a standard pack with all marketing materials unaltered (ST). The study includes a three month purchasing intervention and continued follow-up through 12 months. Throughout the study interactive text messaging assessments will be used to measure acute and persistent impact of labeling and marketing on perceptions of tobacco products, subjective effects of consumption, awareness of tobacco-related harms, tobacco use behavior, and quitting motivation. At three separate time points, participants will: a) complete a web-based questionnaire b) provide a saliva sample for cotinine analysis. The rigorous design and extensive objective measurements are significant innovations on the currently published research in this field and should lead to significant advances in tobacco regulatory science.

DETAILED DESCRIPTION:
Smokers handle their packs frequently. Product packaging is a crucial medium by which the tobacco industry communicates product attributes, including reassurances about risk. The industry uses branded imagery on packs to influence consumer perceptions of their product, while at the same time the tobacco control community uses health warning labels to communicate harmful and potentially harmful constituents and risks of tobacco products. The World Health Organization Framework Convention on Tobacco Control (WHO FCTC) is a treaty enacted to ensure that every person is informed of the health consequences and addictive nature of tobacco consumption. Article 11 of the treaty requires Parties to implement large, rotating health warnings and urges governments to restrict or prohibit the use of Industry logos, colors, brand images or promotional information on packaging other than brand names and product names displayed in a standard color and font style. Study Objective: To conduct a randomized trial of the effect of cigarette pack design on 450 smokers of popular cigarette brands aged 21-65, who are committed to continue smoking (no intention to quit in the next 6-months). These committed smokers will be randomized to have their cigarettes packaged in one of 3 study arms: a) blank pack design with all marketing materials removed (BP), b) blank pack with a large graphic warning label (AM: Australian model) and c) standard pack with marketing materials intact (ST: US model).

ELIGIBILITY:
Inclusion Criteria:

* 21-65 years of age
* A current resident of San Diego County
* Daily smokers of at least 5 cigarettes/day who are classified as in the pre-contemplator stage of change (i.e. do not intend to quit smoking in the next 6-months)
* Regular smokers of popular U.S. cigarette brands
* Have a cell phone with a text messaging service plan

Exclusion Criteria:

* Non-Daily cigarette smokers and daily smokers of alternative brand cigarettes
* Marked organic impairment or unstable medical problems (such as a seizure disorder)
* Current pregnancy or intent to become pregnant during the next 12 weeks
* Prisoners, incarcerated or institutionalized individuals

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Perceptions of Risk From Tobacco Use and Perceptions of Pack Appeal | Assessed over 4-months and 12-months
  Changes in perceptions of risk from tobacco use and appeal of tobacco packs
Changes in Awareness and Concern about Health Hazards | Assessed over 4-months and 12-months
  Changes in perceptions of harm and potential risks
Changes in routinized behavior and persistence over time. | Assessed over 4-months and 12-months
  Decreased willingness to display the pack in public.
Changes in cigarette smoking behaviors. | Assessed over 4-months and 12-months
  Changes in the percent smokers, consumption per smoker, and recent quit attempts validated with saliva cotinine.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Pierce JP, Kealey S, Leas EC, Pulvers K, Stone MD, Oratowski J, Brighton E, Villasenor A, Strong DR. Effect of Graphic Warning Labels on Cigarette Pack-Hiding Behavior Among Smokers: The CASA Randomized Clinical Trial. JAMA Netw Open. 2022 Jun 1;5(6):e2214242. doi: 10.1001/jamanetworkopen.2022.14242. PMID 35653155
- [Derived] Strong DR, Pierce JP, Pulvers K, Stone MD, Villasenor A, Pu M, Dimofte CV, Leas EC, Oratowski J, Brighton E, Hurst S, Kealey S, Chen R, Messer K. Effect of Graphic Warning Labels on Cigarette Packs on US Smokers' Cognitions and Smoking Behavior After 3 Months: A Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2121387. doi: 10.1001/jamanetworkopen.2021.21387. PMID 34347057